CLINICAL TRIAL: NCT03343132
Title: Gait Adaptability: Tracking Locomotor Recovery After Incomplete Spinal Cord Injury Via Sensitive Assessments in a Virtual Reality Treadmill Environment
Brief Title: Gait Adaptability: Tracking Locomotor Recovery After Incomplete Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Foundation Wings For Life (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-01780
Record Dates: First submitted 2017-10-09; First posted 2017-11-17 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Gait Disorders, Neurologic; Gait Disorder, Sensorimotor
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Subacute SCI
  Interventions: Behavioral: Standard locomotor therapy
- Chronic SCI
- Controls

INTERVENTIONS:
Behavioral: Standard locomotor therapy — Typical clinical therapy.
  Groups: Subacute SCI

SUMMARY:
Adaptive gait assessements will be evaluated as a potential new marker for tracking locomotor recovery throughout rehabilitation of spinal cord injury subjects. To this end, controls, subacute and chronic patients will be assessed at two timepoints with 3 month standard rehabilitation inbetween. The specific assessments will require the participant to acitvely modulate their gait pattern to fullfill specific task constraints. Their performance will be assessed via 3D kinematics, kinetics and EMG and these measures will be used to describe the adaptive capacity that the patient retains. Sensitivity and specificity of these markers will be determined. With more sensitive descriptors of gait function and quality, locomotor rehabilitation for SCI can be better designed and smaller effects can be accurately measured.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Healthy controls
* Patients with an incomplete spinal cord injury in a chronic (at least 12 months post-injury) or subacute (3-6 months post-injury) stage of recovery
* Age: 18 years and older
* Able to stand without physical assistance and handrails for more than 120s
* preserved segmental and cutaneo-muscular reflexes in the lower limbs
* Bodyweight over 20 kg and under 120 kg
* Mini-Mental state examination score 26 (test only performed if cognitive deficits are suspected)

Exclusion Criteria:

* Current orthopedic problems
* Neurological impairment other than SCI
* Premorbid major depression or psychosis
* Metal implants in the cervical skull
* History of significant autonomic dysreflexia with treatment
* Dermatological issues (e.g. decubitus) at the harness attachment site (back, abdomen, upper legs)
* Malignant diseases
* Heart insufficiency NYHA III-IV
* Potential pregnancy
* Unlikely to complete the intervention or return for follow-up
* Participation in another training study
* Contraindications for training using the GRAIL (according the manual)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic; community sample
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Change in kinematics | Baseline and through study completion, an average of 4 months
  Recording of movement tasks

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik Balgrist, Zurich, Switzerland

REFERENCES:
- [Derived] Zipser-Mohammadzada F, Scheffers MF, Conway BA, Halliday DM, Zipser CM, Curt A, Schubert M. Intramuscular coherence enables robust assessment of modulated supra-spinal input in human gait: an inter-dependence study of visual task and walking speed. Exp Brain Res. 2023 Jun;241(6):1675-1689. doi: 10.1007/s00221-023-06635-4. Epub 2023 May 18. PMID 37199775
- [Derived] Mohammadzada F, Zipser CM, Easthope CA, Halliday DM, Conway BA, Curt A, Schubert M. Mind your step: Target walking task reveals gait disturbance in individuals with incomplete spinal cord injury. J Neuroeng Rehabil. 2022 Mar 25;19(1):36. doi: 10.1186/s12984-022-01013-7. PMID 35337335